CLINICAL TRIAL: NCT03211598
Title: Pilot Trial Assessing the Technical Feasibility and Safety of the Surefire Infusion System for Use in DEB-TACE (Surefire)
Brief Title: Surefire Institutional DEB-TACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexander Kim (Other)
Collaborators: Surefire Medical, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Alexander Kim, Chief of Interventional Radiology at Medstar Georgetown University Hospital, Georgetown University
Organization: Georgetown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SF Georgetown
Record Dates: First submitted 2017-03-21; First posted 2017-07-07 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE with Surefire (Other): Subjects enrolled in the study will have their TACE procedure with the Surefire Infusion System.
  Interventions: Procedure: TACE with Surefire

INTERVENTIONS:
Procedure: TACE with Surefire — Subjects that consent to the study will receive their TACE procedure through the Surefire Infusion System

SUMMARY:
The purpose of this study is to determine the feasibility and safety of the Surefire Infusion System (SIS) for delivery of Drug Eluting Beads Transcatheter Chemoembolization (DEB-TACE) in the HCC population. This study will allow us to determine the effectiveness of SIS for HCC in terms of disease response.

DETAILED DESCRIPTION:
This is a single arm pilot study to evaluate the technical feasibility and safety of performing DEB-TACE using the investigational delivery device: Surefire Infusion System (SIS). Patients presenting with primary liver cancer without evidence of metastatic disease or vascular invasion will be considered for the trial. Patients enrolled in the trial will undergo 1 or 2 sessions of DEB-TACE delivered through SIS as determined by the performing interventional radiologist. Decision for second treatment will be based on the degree of disease burden and vascular anatomy demonstrated on the first treatment session. To limit potential hepatotoxicity, patients with multifocal disease in a single lobe may be treated with a 2nd treatment with the investigational device. Patients with a large lesion being supplied by multiple vessels may also undergo a 2nd treatment session based on the investigator's judgement. The decision to proceed with a second treatment will be determined at the time of the first treatment based on disease burden and vascular anatomy. There will be an interval of 2-4 weeks between treatments. All patients undergoing 2nd treatment will have a repeat laboratory evaluation with treatment deferred for 2-4 weeks for those not meeting initial inclusion criteria. For patients who labs have not normalized at this time will not undergo a 2nd treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Primary liver cancers based on biopsy or imaging criteria
2. Child-Pugh A or B7 liver disease
3. Bilirubin <2.0 mg/dL
4. Albumin >3.0 gm/dL
5. ECOG status 0 or 1
6. Adequate renal function

   a. Creatinine < 2.0 mg/dL
7. Age 18 or older
8. Able to understand informed consent
9. Life expectancy > 3 months
10. Women of childbearing potential must have a negative serum/urine pregnancy test on the day of planned procedure.

Exclusion Criteria:

1. Portal vein thrombus
2. Uncontrolled ascites
3. Hepatic encephalopathy
4. Uncorrectable coagulopathy (platelets <50,000, INR >1.50)
5. Untreatable contrast allergy
6. Pregnancy
7. Symptomatic congestive heart failure
8. Prior systematic therapy for HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Stasis of flow in target vessel as seen on digital subtraction angiography or cone-beam CT, or reflux of particles despite the use of SIS. | During chemoembolization
  Assess the technical feasibility of performing TACE using the SIS. If stasis of flow is not reached after 1 vial of DEB, further bland embolization will be performed until stasis is reached or earlier as determined adequate by the treating interventional radiologist.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Duration of study (12 months)
  Assess the safety of SIS for TACE as per CTCAE v 4.03

SECONDARY OUTCOMES:
Tumor Assessment via MRI Imaging | Duration of study (12 months)
  Assess the disease response rates of HCC with TACE using the SIS per mRECIST criteria
Tumor Assessment via CT Imaging | Duration of study (12 months)
  Assess the disease response rates of HCC with TACE using the SIS per mRECIST criteria
FACT Hep4 Questionnaire | Visit 5 (week 5)
  Correlate outcomes with treatment endpoint, defined as stasis of flow in target vessel on DSA or CBCT, or reflux of particles despite the use of SIS

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Y Kim, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee KK, Kim DG, Moon IS, Lee MD, Park JH. Liver transplantation versus liver resection for the treatment of hepatocellular carcinoma. J Surg Oncol. 2010 Jan 1;101(1):47-53. doi: 10.1002/jso.21415. PMID 19798686